CLINICAL TRIAL: NCT05516095
Title: The Antidepressant Effect of Intermittent Theta Burst Stimulation (iTBS) A Randomised Double-blind Sham-controlled Trial
Brief Title: The Antidepressant Effect of Intermittent Theta Burst Stimulation (iTBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 228765; HNF1578-21 (Other Grant/Funding Number: Northern Norway Regional Health Authorithy)
Record Dates: First submitted 2022-02-14; First posted 2022-08-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2022-06

CONDITIONS: Depression; Executive Dysfunction
Keywords: moderate depression; major depression
MeSH Terms: conditions — Depression; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Randomized placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization will be performed in MatLab (https://se.mathworks.com/products/matlab.html), with the "randperm" command that perform randomization in four permuted blocks to groups and gender in a single operation. The randomization procedure in MatLab will be performed by the Research Department at the University Hospital North-Norway, and they will produce numbered colored envelopes (e.g. pink = female, blue = male) containing number of the coil (e.g. 1= active, 2 = sham) that will be opened by the research assistant who mount the coil before the clinician start the treatment procedure. Thus, neither the clinician nor the patient will know which treatment that is provided, but the patient will be asked to guess their group allocation at the follow-up four weeks after the treatment end, as recommended in recent repetitive transcranial magnetic stimulation (rTMS) guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active iTBS (Active Comparator): iTBS will be delivered with 120% of resting motor threshold, triplet 50 Hz bursts repeated at 5 Hz; 2 seconds on and 8 s off, 600 pulses per session with a total duration of 3 min 9 s. Treatment will be provided for 10 days for two consecutive weeks (except Saturdays and Sundays). Each patient will start treatment at the same time between 9 am and 3 pm during the 10-day treatment period.
  Interventions: Device: Transcranial magnet stimulation
- Sham iTBS (Placebo Comparator): The sham system has an identical look, weight and sound compared to the true coil, and delivers electrical stimulation that can be felt at the skin but without penetrating the skull and thus not inducing any treatment effect. The sham stimulation will be given with the same procedure as the active stimulation; 2 seconds on and 8 s off, 600 pulses per session with a total duration of 3 min 9 s.
  Interventions: Device: Sham Transcranial magnet stimulation

INTERVENTIONS:
Device: Transcranial magnet stimulation — Theta burst stimulation, which is a form of Transcranial magnet stimulation, works by inducing focused magnetic field pulses to make durable changes in the activity of brain regions. The magnetic pulses are transferred to the brain through an electromagnetic coil.
  Other Names: Theta burst stimulation
  Arms: Active iTBS
Device: Sham Transcranial magnet stimulation — Similar in appearance and give the same sound as the active device, but deliver no magnetic pulse that reach the brain
  Other Names: Sham Theta burst stimulation
  Arms: Sham iTBS

SUMMARY:
The present study is a randomized placebo-controlled trial examining the effect of intermittent theta burst stimulation (iTBS) on unipolar depression. iTBS is a form of transcranial magnet stimulation.

The anti-depressive effect of two weeks of once- a - day neuronavigated iTBS over the dorsolateral left prefrontal cortex (DLPFC) will be investigated in comparison to sham (placebo) iTBS. Previous studies have shown that iTBS is an effective treatment for reducing symptoms of depression, but it is still unclear why some patients have a strong response to iTBS, whereas others show less or no reduction to test possible factors that can explain the inter-individual response to iTBS.

Measures of cognitive functions, structural and functional brain data measured by Magnetic Resonance imaging (MRi), quality of life, sleep quality, general health status, and genetic measures will be obtained to answer the goals of this study.

The main hypotheses are: 1) Patients receiving iTBS will display significantly larger reductions in depressive symptoms measured by the Montgomery-Asberg Depression Rating Scale and Becks Depression Inventory II compared to patients receiving sham stimulation. 2) Reduction in depressive symptoms will be significantly associated with a concomitant improvement in executive functions measured by neuropsychological tests. 3) Stronger connectivity at baseline between the DLFPC and the anterior cingulate cortices will be associated with better response to iTBS. 4) Variability in genetic measures will be significantly associated with treatment response to iTBS. 5) Variability in white matter structural measures of the brain will be significantly associated with the anti-depressive response to iTBS.

Participants will be recruited prospectively, and the study performed at a single university hospital. After written informed consent is obtained from eligible, volunteering patients, baseline measurements will be administrated, and the patient will be allocated to either sham or active iTBS once a day for 10 consecutive workdays. Four weeks after the last treatment day, the patients will be followed up by phone interviews.

ELIGIBILITY:
Inclusion Criteria:

* A MADRS score of =/ > 20 (moderate depression).
* The current depressive episode must have lasted more than 2 weeks but less than 2 years
* Drug therapy must have been stable for the last three weeks prior to the first treatment day with iTBS and is to be kept stable throughout the study until 4 weeks after the last day of iTBS treatment.
* Patients must volunteer to provide informed consent, be able to follow the treatment schedule and have a satisfactory safety screening for iTBS and MRI.

Exclusion Criteria:

* The current depressive episode is in the mild range or contrary that the current episode fulfills the criteria for a major depressive episode requiring inpatient treatment and/or electroconvulsive therapy.
* The current depressive episode is clearly triggered by grief or a recent major stressful life event.
* Bipolar disorder.
* Borderline personality disorder.
* Psychotic symptoms the last 6 months.
* Alcohol or substance abuse/addiction in the last 6 months.
* Current eating disorders.
* Obsessive- compulsive disorders.
* Post-traumatic stress disorder.
* Any medical history of seizure.
* Any neurological or neurosurgical pathologies.
* Any current cardiac or systemic disease.
* Metallic prosthetic material or foreign objects in the body (pacemakers, internal cardioverter defibrillator units, insulin pump, prosthetic eye equipment, etc.).
* Previously diagnosed developmental disorder.
* Pregnancy or lactating.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale. | Up to 4 months.
  Clinician rated depression inventory.
Beck's Depression Inventory - II. | Up to 4 months.
  Patient reported depression inventory.

SECONDARY OUTCOMES:
Beck's Anxiety Inventory. | Up to 4 months.
  Patient reported anxiety inventory.
Wisconsin Card Sorting Test. | Up to 2 weeks.
  Performance based measure of executive functions.
Delis-Kaplan Executive Function System. | Up to 2 weeks.
  Performance based measure of executive functions.
Brief-A | Up to 4 months.
  Questionnaire for self-reported executive functioning.
Whodas 2.0 | Up to 4 months.
  Self-reported disability assessment schedule.
Pittsburgh Sleep Quality Index. | Up to 4 months.
  Self-reported measure of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Aslaksen, PhD, Principal Investigator — UiT The Arctic University of Norway; Marte C Ørbo, PhD, Principal Investigator — UiT The Arctic University of Norway; Ole Grønli, MD, PhD, Principal Investigator — University Hospital North Norway
Locations (1):
- University Hospital North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for outcome measures in the study.
Supporting Information: SAP, Analytic Code
Time Frame: Data used for publications in peer-reviewed journals will be shared after publication at the open data platform used at UiT the Arctic University of Norway.
Access Criteria: Open for everyone.
URL: https://dataverse.no/dataverse/uit

REFERENCES:
- [Derived] Orbo MC, Gronli OK, Larsen C, Vangberg TR, Friborg O, Turi Z, Mittner M, Csifcsak G, Aslaksen PM. The antidepressant effect of intermittent theta burst stimulation (iTBS): study protocol for a randomized double-blind sham-controlled trial. Trials. 2023 Oct 2;24(1):627. doi: 10.1186/s13063-023-07674-6. PMID 37784199